CLINICAL TRIAL: NCT01308996
Title: A Prospective, Open Label, Randomized, Multicenter, Controlled Clinical Study of INFUSE® Bone Graft Used as an Alternative to Autogenous Bone Graft for Vertical Alveolar Ridge Augmentation
Brief Title: Clinical Study of INFUSE® Bone Graft Compared to Autogenous Bone Graft for Vertical Ridge Augmentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Collaborators: Averion International Corporation (Industry); Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G100313
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2012-08

CONDITIONS: Alveolar Bone Loss in Mandible; Edentulous Alveolar Ridge In Mandible
Keywords: alveolar ridge augmentation; edentulous ridge; alveolar ridge defect; posterior mandible defect; bone morphogenic protein; osseointegration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INFUSE® Bone Graft (Experimental)
  Interventions: Device: INFUSE® Bone Graft
- Autogenous bone graft (Active Comparator)
  Interventions: Procedure: Autogenous bone graft from tibia or iliac crest

INTERVENTIONS:
Device: INFUSE® Bone Graft — Implantation of INFUSE® Bone Graft [recombinant human Bone Morphogenetic Protein-2 (rhBMP-2)] and absorbable collagen sponge (ACS) carrier at 1.50 mg/cc with space maintenance device
  Arms: INFUSE® Bone Graft
Procedure: Autogenous bone graft from tibia or iliac crest — Implantation of autogenous bone graft from iliac crest or tibia with titanium mesh space maintenance device
  Arms: Autogenous bone graft

SUMMARY:
The purpose of this study is to evaluate the INFUSE® Bone Graft as an alternative to autograft for bone formation in the back of the mandible (lower jaw) prior to placing dental implants.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate INFUSE® Bone Graft as an alternative to autograft for alveolar ridge bone formation in the posterior mandible prior to dental implants. A subject must have a defect behind the canine of 2-4 teeth for at least 2 months and be a candidate for dental implants.

ELIGIBILITY:
Inclusion Criteria:

1. Has been edentulous for at least 2 months with an alveolar ridge defect affecting 2-4 teeth in the posterior mandible, posterior to the canine.
2. Has an alveolar ridge defect with a minimum starting height of 5 mm above the superior cortex of the inferior alveolar canal in the posterior mandible.
3. Is a candidate for dental implants (2-4 teeth) in the affected posterior mandibular alveolar ridge area.
4. Has a prosthodontic treatment plan in place.
5. Has no known condition that would interfere with collecting autogenous bone at either the tibia or the iliac crest for a bone grafting procedure.
6. Is 21-75 years of age (inclusive).
7. If female of childbearing potential, has a negative urine pregnancy test, is not lactating, and agrees not to become pregnant for at least 12 months after surgery.
8. Is able to comply with all study-related procedures, including exercising good oral hygiene.
9. Is able to provide written informed consent.

Exclusion Criteria:

1. Has bilateral alveolar ridge defects requiring simultaneous augmentation or a second augmentation planned during the course of the study.
2. Has an active infection at the planned augmentation site.
3. Has active periodontal disease of Grade III or higher.
4. Has had a dental extraction procedure at the planned augmentation site within the 2 months prior to Day 0.
5. Has had a soft tissue graft at the planned augmentation site within less than 2 weeks of Screening.
6. Is expected to require any additional bone graft material (e.g., allograft and xenograft) at the planned augmentation site in addition to the investigative treatment or autogenous bone, as determined by the investigator prior to surgery.
7. Has a history of a failed alveolar ridge augmentation procedure.
8. Has a pathology finding that would either compromise a bone grafting procedure or interfere with obtaining quantitative measurements from postoperative CT scans.
9. Is an insulin-dependent diabetic.
10. Has an overt or active systemic infection, such as human immunodeficiency virus (HIV), bacteremia, or hepatitis C virus (HCV).
11. Has a planned augmentation site in the area of a resected or extant tumor.
12. Has presence of an active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
13. Is actively using any nicotine-containing products such as, but not limited to, smoking and chewing tobacco, nicotine patch, nicotine gum, etc. within 2 weeks prior to Screening.
14. Is alcohol or drug dependent, as determined by the investigator.
15. Is taking medications or having treatment known to have an effect on bone metabolism, such as, but not limited to:

    * calcitonin within the past 6 months;
    * fluorides for 30 days or more within the past 12 months;
    * cumulative use of oral bisphosphonates for less than 5 years within the past 6 months;
    * cumulative use of oral bisphosphonates for 5 years or more;
    * any previous use of intravenous bisphosphonates;
    * chronic tetracycline (e.g., ongoing within the past month) or tetracycline analogs within the past 12 months;
    * estrogen replacement therapy within the past 2 months; or
    * methotrexate within the past 12 months.
16. Has a disease that affects bone metabolism, such as:

    * congenital connective tissue disease (e.g., Ehlers-Danlos syndrome, osteogenesis imperfecta);
    * hyperthyroidism; or
    * hyperparathyroidism.
17. Has a history of autoimmune disease (e.g., systemic lupus erythematosus, dermatomyositis, rheumatoid arthritis, etc.).
18. Has any previous exposure to any recombinant BMPs of either human or animal extraction.
19. Has a known history of prior exposure to silicone or injectable collagen implants.
20. Has a known hypersensitivity or allergy to collagen or protein pharmaceuticals (e.g., monoclonal antibodies or gamma globulins).
21. Has a known hypersensitivity or allergy to titanium.
22. Has a history of allergy to bovine collagen products.
23. Has chronic or acute renal failure
24. Has chronic or acute liver failure.
25. Has received treatment with an investigational therapy (drug, device, and/or biologic) within 30 days prior to bone graft implantation surgery or such treatment is planned during the 12-month period following the study surgery.
26. Has any condition that in the judgment of the investigator would place the subject at undue risk or interfere with the results of the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Osseous volumetric fill underneath the titanium mesh of edentulous sites in the posterior mandible. | 210 days

SECONDARY OUTCOMES:
Pain level at the surgical site, as well as at the donor site (if applicable). | 210 days
  Numerical rating scales used to evaluate pain intensity and frequency.
Ability to place dental implants | 210 days
Histological evaluation (percent vital bone) | 210 days
Surgical failure rate | 210 days
Adverse Events | 210 Days